CLINICAL TRIAL: NCT06941168
Title: Potential Advantages of Robotic Total Gastrectomy in Advanced Middle-Upper Gastric Cancer
Brief Title: Potential Advantages of Robotic Total Gastrectomy in Advanced Middle-Upper Gastric Cancer: A Multicenter Propensity Score Matching Analysis
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Chief of Gastric Cancer Surgery, Fujian Medical University
Other Study IDs: FJMU0416
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Advanced Gastric Cancer
Keywords: Robotic surgery; advanced middle-upper gastric cancer; Total gastrectomy; Perioperative outcomes; Oncologic outcomes
MeSH Terms: interventions — ezogabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RTG: Patients who underwent robotic total gastrectomy
  Interventions: Procedure: Robotic Total Gastrectomy and Laparoscopic Total Gastrectomy
- LTG: Patients who underwent laparoscopic total gastrectomy
  Interventions: Procedure: Robotic Total Gastrectomy and Laparoscopic Total Gastrectomy

INTERVENTIONS:
Procedure: Robotic Total Gastrectomy and Laparoscopic Total Gastrectomy — RTG:Robotic total gastrectomy with D2 lymphadenectomy performed using the Da Vinci Surgical System, following the Japanese Gastric Cancer Treatment Guidelines.
  LTG:Laparoscopic total gastrectomy with D2 lymphadenectomy performed by experienced surgeons following standardized procedures, based on the Japanese Gastric Cancer Treatment Guidelines.
  Other Names: RTG and LTG

SUMMARY:
This multicenter retrospective cohort study aimed to evaluate the potential advantages of robotic total gastrectomy (RTG) compared to laparoscopic total gastrectomy (LTG) in patients with advanced middle and upper gastric cancer (AMUGC). A total of 1,099 patients who underwent radical total gastrectomy between 2013 and 2020 were included. After strict inclusion and exclusion criteria, propensity score matching (1:1) was conducted to balance baseline characteristics. The primary endpoint was 3-year disease-free survival (DFS), with secondary outcomes including overall survival, recurrence rates and patterns, and perioperative outcomes. All procedures were performed by experienced surgeons following standardized protocols across eight high-volume centers. Data quality was ensured through a centralized electronic system, unified training, and rigorous verification. This study provides real-world evidence on surgical outcomes and long-term prognosis, contributing to clinical decision-making in the treatment of AMUGC.

DETAILED DESCRIPTION:
All patients provided informed consent for the use of their clinical data at admission or prior to surgery, in accordance with the Declaration of Helsinki. The study protocol was approved by the institutional review boards of all eight participating centers and reported in accordance with STROCSS guidelines.

This multicenter registry included patients diagnosed with middle and upper gastric cancer (GC), who underwent radical total gastrectomy with pathological staging of T2-4aN0-3bM0. Exclusion criteria included ASA class >3, residual GC, neoadjuvant chemotherapy, combined organ resection, indocyanine green (ICG) use, concurrent/past malignancies, and loss to follow-up. A total of 1,099 eligible patients were included in the final analysis, with 237 receiving robotic total gastrectomy (RTG) and 862 receiving laparoscopic total gastrectomy (LTG).

To ensure surgical quality, all centers followed standardized protocols. Surgeons had completed their institutional learning curve-defined as independently performing ≥50 laparoscopic gastrectomies with consistent outcomes-before enrolling patients. RTG was performed only by certified surgeons trained in the Da Vinci Robotic System. Surgical procedures adhered to Japanese Gastric Cancer Treatment Guidelines, and pathological staging followed the AJCC 8th edition criteria. Resected specimens were evaluated by experienced gastrointestinal pathologists using uniform histopathological protocols. R1 resection was defined as microscopic tumor presence at the surgical margin.

Patient selection for RTG or LTG was based on shared decision-making, considering tumor stage, comorbidities, surgical risk, cost, and patient preference. Informed consent included agreement to cover any additional costs associated with robotic surgery.

Propensity score matching (PSM) was used to control for baseline differences between groups. A 1:1 nearest-neighbor matching with a caliper of 0.2 was performed using the MatchIt package in R. Thirteen covariates-age, sex, BMI, ASA grade, comorbidities, tumor size/location, histology, pT/pN stage, lymphadenectomy extent, adjuvant chemotherapy, and year of surgery-were included. Matching balance was evaluated using standardized mean differences (SMDs), with <0.1 considered acceptable.

The registry incorporated a structured follow-up system. Patients were followed every 3-6 months in the first two years, every 6-12 months between years 3-5, and annually thereafter. Follow-up assessments included physical exams, lab tests, imaging (X-ray, ultrasound, or CT), and annual endoscopy. Telephone follow-up was used to supplement outpatient visits. Recurrence was confirmed through clinical history, imaging, and pathology (preferably biopsy).

Data integrity was ensured through multiple layers of quality control. All participating centers used a standardized electronic data capture (EDC) system. Data entry was performed by trained personnel and verified by designated staff. Regular audits, backtracking of missing data, and cross-checking by two independent researchers were conducted before data export. These procedures ensured accuracy, completeness, and consistency of the registry data.

Statistical analyses were performed using SPSS v26.0 and R v4.4.1. Continuous variables were analyzed via t-tests or Mann-Whitney U tests; categorical variables via chi-square or Fisher's exact tests. Survival was assessed using Kaplan-Meier and Cox regression models, with competing risk models used for recurrence. All tests were two-sided, with a significance level of P<0.05.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with middle or upper gastric cancer (GC)

Pathological stage T2-T4a, N0-N3b, M0 (postoperative)

Underwent radical total gastrectomy

Exclusion Criteria:

- American Society of Anesthesiologists (ASA) class > 3

Residual gastric cancer

Use of indocyanine green (ICG) during surgery

Received neoadjuvant chemotherapy

History of concurrent or previous malignancies

Combined resection of other organs

Lost to follow-up

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with middle or upper gastric cancer who underwent radical total gastrectomy at one of eight high-volume surgical centers in China between 2015 and 2019. Eligible patients had pathologically confirmed stage T2-4aNO-3bмоdisease, with no history of neoadjuvant therapy or other malignancies. All patients were treated according to standardized surgical and pathological protocols and had complete follow-up data for postoperative outcomes and survival analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1099 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2024-08 (Actual)

PRIMARY OUTCOMES:
3-year Disease-Free Survival (DFS) | 3 years after surgery
  Disease-free survival was defined as the time between the date of surgery and date of the last follow-up for recurrence, death, or no recurrence

SECONDARY OUTCOMES:
3-year overall survival (OS) | 3 years after surgery
  Overall survival was defined as the time from the date of surgery to death or last follow-up
3-year Cumulative Incidence of Recurrence (CIR) | 3 years after surgery
  The cumulative incidence of recurrence, including local recurrence, peritoneal, liver, multiple, or other metastatic sites. Competing risk model is used with death from other causes as a competing event.
Recurrence Patterns | Up to 3 years after surgery
  First recurrence location classified as local, peritoneal, hepatic, multiple-site, or other/unspecified. Determined via imaging, pathology during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastric Surgery， Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No